CLINICAL TRIAL: NCT03419741
Title: Repetitive Transcranial Magnetic Stimulation For Smoking Cessation In Cancer Patients
Brief Title: Brain Stimulation For Cancer Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00066330
Record Dates: First submitted 2018-01-02; First posted 2018-02-05 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-04

CONDITIONS: Cancer of Head and Neck; Breast Cancer; Prostate Cancer; Nicotine Dependence
Keywords: Cancer, Nicotine Addiction, Smoking Cessation
MeSH Terms: conditions — Head and Neck Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Tobacco Use Disorder; Neoplasms; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded design of active rTMS and sham rTMS. The pilot will include a total of 20 nicotine-dependent patients with cancer. Subjects will be randomized to either sham rTMS or real rTMS over the left DLPFC. At the end of 7-day study, everyone can be referred to the Hollings Cancer Center (HCC) Tobacco Treatment Program for active treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham TMS
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active rTMS treatment (Active Comparator): Transcranial Magnetic Stimulation Clinical Research System will be used for the active rTMS treatment. Stimulation frequency for all active subjects: 10 Hertz - Pulse train duration (on time) 5 seconds, Inter-train interval (off time) 10 seconds (15 second cycle time), Power (intensity) level 100% resting motor threshold, Total 60 trains, 15 minutes, Total pulses 3000 per day, 3000 x 5 = 15000 pulses for 5 sessions.
  Interventions: Device: Transcranial Magnetic Stimulation Clinical Research System
- Sham rTMS treatment (Sham Comparator): Transcranial Magnetic Stimulation Clinical Research System -sham TMS will be connected to an electrical generator on a 9 V battery and electrodes will be placed over the prefrontal cortex. The regulator is triggered by the TMS machine to allow brief, microsecond, pulses of the electrical current through to the skin on the subjects' forehead. Electrical stimulation will be triggered by the TMS machine to correspond to the sham TMS pulses.
  Interventions: Device: Transcranial Magnetic Stimulation Clinical Research System

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation Clinical Research System — Transcranial Magnetic Stimulation Clinical Research System is a US FDA approved treatment system for depression. The treatment research system includes motor threshold TMS coil, active TMS coil and sham TMS coil.

SUMMARY:
Smoking cessation and relapse prevention represent and important opportunity to improve cancer survival rates, reduce the risk of cancer treatment complication, and improve the quality of life of patients with and survivors of cancer. Previous studies showed that repetitive TMS (rTMS) reduced cue craving to smoking and treat nicotine dependent smokers. Recently one study completed by our team demonstrated that 10 sessions of rTMS over the left dorsolateral prefrontal cortex (DLPFC) reduced cigarette consumption and cue craving, and also increased quitting rate on target quit date in nicotine dependent smokers. Thus, we propose conducting a controlled, double-blind trial comparing the effect of treatments of active rTMS and sham rTMS on cigarette abstinence days, cigarette consumption and smoking craving during a 7-days of quit attempt period in 20 nicotine-dependent patients with cancer. Specific aims are: Aim 1: Assess a feasibility of the rTMS for smoking cessation in cancer patients. Aim 2: Obtain preliminary estimates of whether one-week active rTMS of left DLPFC tends to be more efficacious than sham rTMS during a 7-days of quit attempt laboratory model period increasing abstinence days, and also decreasing cigarette consumption and cue-elicited craving in cancer patients with smoking.

DETAILED DESCRIPTION:
Specific aims: Smoking cessation and relapse prevention represent and important opportunity to improve cancer survival rates , reduce the risk of cancer treatment complication, and improve the quality of life of patients with and survivors of cancer . Previous studies showed that repetitive TMS (rTMS) reduced cue craving to smoking and treat nicotine dependent smokers. Recently one study completed by our team demonstrated that 10 sessions of rTMS over the left dorsolateral prefrontal cortex (DLPFC) reduced cigarette consumption and cue craving, and also increased quitting rate on target quit date in nicotine dependent smokers. Thus, we propose conducting a controlled, double-blind trial comparing the effect of treatments of active rTMS and sham rTMS on cigarette abstinence days, cigarette consumption and smoking craving during a 7-days of quit attempt period in 20 nicotine-dependent patients with cancer. Specific aims are: Aim 1: Assess a feasibility of the rTMS for smoking cessation in cancer patients. Aim 2: Obtain preliminary estimates of whether one-week active rTMS of left DLPFC tends to be more efficacious than sham rTMS during a 7-days of quit attempt laboratory model period increasing abstinence days, and also decreasing cigarette consumption and cue-elicited craving in cancer patients with smoking.

1.1. Primary objective To assess a feasibility of the rTMS for smoking cessation in cancer patients: The primary feasibility measures are : whether or not we can enroll 20 cancer patients with smoking within 12 months? 1.2 Secondary objectives

(1) Study attrition. How many subjects can complete 7-day quit attempt during rTMS treatment? How many subjects will complete one-month follow-up? (2) To obtain preliminary estimates of whether one-week active rTMS of left DLPFC tends to be more efficacious than sham rTMS during a 7-days of quit attempt laboratory model period increasing abstinence days, and also decreasing cigarette consumption and cue-elicited craving in cancer patients with smoking.

1.3 Exploratory objectives Self-reported number of cigarettes smoked per day, The brief questionnaire of smoking urges (QSU - Brief), visual analog scale for craving and side effect will be measured pre and post each rTMS session. Other assessment, Carbon Monoxide, Fagerstrom Test for Nicotine Dependence (FTND), and Minnesota Nicotine withdrawing Scale (MNWS) will be completed at baseline and the last TMS. Quitting attempt will verify daily CO < 5 ppm. FTND, Feasibility metrics will also be tracked, including numbers of complete TMS sessions and dropout rate.

ELIGIBILITY:
Inclusion Criteria:

* 1. Completed cancer treatment (e.g. surgery, chemotherapy and radiation) > 6 months Patients with current endocrine therapy will be included for the study.

  2. Have been diagnosed with noninvasive or invasive (Stage 1, 2, or 3A) breast cancer or prostate cancer.

  3. Smoke 5 or more cigarettes per day and have a carbon monoxide (CO) level > 5 ppm indicative of recent smoking.

  4. Not have received substance abuse treatment within the previous 30 days. 5. Meet criteria for low to moderate nicotine dependence as determined by FTND ≥1.

  6. Be willing to provide informed consent. 7. Be able to comply with protocol requirements and likely to complete all study procedures.

  8. Is willing to consider trying to quit smoking. 9. Have no active cardiac, neurologic, or psychiatric illness. 10. 0.5-10 years post diagnosis of cancer at the time enrollment.

Exclusion Criteria:

1. Current dependence, defined by Diagnostic and Statistical manual of Mental Disorders (DSM)-V criteria, on any psychoactive substances other than nicotine or caffeine.
2. Contraindication to rTMS (history of neurological disorder or seizure, increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for > 15 minutes, implanted electronic device, metal in the head, or pregnancy).
3. History of autoimmune, endocrine, viral, or vascular disorder affecting the brain.
4. History of neurological disorder that would lead to local or diffuse brain lesions or significant physical impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-21 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Li X, Hartwell KJ, Owens M, Lematty T, Borckardt JJ, Hanlon CA, Brady KT, George MS. Repetitive transcranial magnetic stimulation of the dorsolateral prefrontal cortex reduces nicotine cue craving. Biol Psychiatry. 2013 Apr 15;73(8):714-20. doi: 10.1016/j.biopsych.2013.01.003. Epub 2013 Feb 26. PMID 23485014

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active rTMS Treatment | Sham rTMS Treatment
Started | 5 | 6
Treated (Treated: to indicate the number of participants who began treatment.) | 4 | 4
Completed | 3 | 4
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: 13 were invited for a screening visit, 11 met study criteria, all of whom enrolled. Three participants declined before treatment initiation. Eight participants were randomized and started the treatment. Among the 8 participants who started treatment, 4 received sham treatment and the other 4 received active rTMS treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS Treatment | Sham rTMS Treatment | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] | 63.25 [60 to 66] | 64.5 [60 to 68] | 63.9 [60 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Three participants did not show up for treatment.
  Participants
    number analyzed (Participants) | 4 | 4 | 8
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 4 | 3 | 7
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Cigarette per day = the number of smoked cigarettes per 24 hours [Mean (Full Range); unit: cigarettes] | 15 [6 to 30] | 10 [6 to 20] | 13 [6 to 30]

OUTCOME MEASURES:

1. Primary Outcome: The Number of Enrollment
Description: How many cancer patients with smoking can be enrolled in 12 months?
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Active rTMS Treatment | Sham rTMS Treatment
Number analyzed (Participants) | 4 | 4
participants | 4 | 4
Statistical Analysis 1: Comparison: Active rTMS Treatment vs Sham rTMS Treatment; Test type: Other — We plan to enroll 20 participants within one year. Eleven participants were enrolled. 11/20 = 55% completed the number of enrollment; percentage; % = 11

2. Secondary Outcome: Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) on the Number of Abstinence Days.
Description: Total number of smoke-free days during a day quit attempt. Self-reported abstinence during the day quit attempt will be assessed via timeline. The maximum number of consecutive days of abstinence will be recorded. Participants who does not report at least one 24-hour period of abstinence will be recorded as "0" days abstinent.
Time Frame: 5 days
Measure: Number; unit: days
Arm/Group | Active rTMS Treatment | Sham rTMS Treatment
Number analyzed (Participants) | 4 | 4
days | 0 | 0

3. Other Pre Specified Outcome: Effect of rTMS on Cigarette Consumption
Description: the change of self-reported number of cigarettes smoked per day
Time Frame: 5 days
Measure: Mean (Standard Error); unit: number of cigarettes
Arm/Group | Active rTMS Treatment | Sham rTMS Treatment
Number analyzed (Participants) | 3 | 4
number of cigarettes | 12.17 (1.48) | 11.29 (1.71)

4. Other Pre Specified Outcome: Effect of rTMS on Cue Craving to Smoke Cigarette
Description: Brief questionnaire of smoking urges - brief (QSU - Brief) is used to assess smoking urges. Ten questions are included in the test. Range of scales is 1-7 score for each item. The cue craving scales include 10 items. The range of the total score is 10- 70 score. The maximum number means the highest craving that is the worst outcome. The minimum number is the least craving for cigarettes that is the best outcome.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS Treatment | Sham rTMS Treatment
Number analyzed (Participants) | 3 | 4
score on a scale
  Session 1 | 45.3 (24.9) | 36.0 (43.7)
  Session 5 | 25.6 (24.1) | 32.8 (44.7)

5. Other Pre Specified Outcome: Effect of rTMS on Cue Craving to Smoke Cigarette
Description: The change of visual analog scale (VAS). The VAS has 1-7 score. The minimum is 1 which means the best result. The maximum value of 7 is the worst outcome. The VAS was measured during 5 treatment sessions.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS Treatment | Sham rTMS Treatment
Number analyzed (Participants) | 3 | 4
score on a scale
  Session 1 | 5.2 (2.1) | 3.8 (2.9)
  Session 5 | 3.7 (3.2) | 3.5 (3.1)

6. Other Pre Specified Outcome: Adverse Events
Description: Side effect will be measured pre and post each rTMS session.
Time Frame: 5 days
Measure: Number; unit: number of events
Arm/Group | Active rTMS Treatment | Sham rTMS Treatment
Number analyzed (Participants) | 4 | 4
number of events | 2 | 0

7. Other Pre Specified Outcome: Study Attrition Rate
Description: How many subjects completed treatment and a 30 days follow-up.
Time Frame: 12 months
Population: One dropped out of the study.
Measure: Number; unit: participants
Arm/Group | Active rTMS Treatment | Sham rTMS Treatment
Number analyzed (Participants) | 4 | 4
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data will be collected throughout the course of the treatment part of the study, up to 30 days. We estimated adverse events through study completion, an average of 30 days.
Description: Adverse events include headache and pain on the stimulation site.
Arm/Group | Active rTMS Treatment | Sham rTMS Treatment
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS Treatment (N=4) | Sham rTMS Treatment (N=4)
confusional state (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — The participant showed a confusional state, disorientation, and difficulty following commands. The PI detected the SAE during the pre-session assessment and was thus deemed not to be related to TMS treatment. The confusion resulted from hypoxemia.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS Treatment (N=4) | Sham rTMS Treatment (N=4)
taste change (Nervous system disorders) | 1 (1) | 0 (0) — One participant reported a metalic taste after active TMS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT03419741/Prot_SAP_000.pdf